CLINICAL TRIAL: NCT00586417
Title: A Research Pilot Study in Healthy Volunteers to Evaluate Biomarkers for Novel Anticancer Treatments.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00012830
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: angiogenesis; tumor angiogenesis; biomarkers; healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This is a basic research study. There are no treatments with drugs or devices. Wound healing is being studied in healthy volunteers.
  Interventions: Other: punch biopsy

INTERVENTIONS:
Other: punch biopsy — skin biopsies

SUMMARY:
The overall goal of this study is to determine the feasibility and the variability of several biomarker assays in normal subjects that are relevant to tumor biology and novel anti-cancer treatments, with the goal of refining these assays for use in future therapeutic studies.

DETAILED DESCRIPTION:
Many physiological processes in normal growth, development, injury, and repair are critical for tumor growth and progression. Usually these processes are deregulated, allowing for the potential of tumor selectivity in targeting many of these processes. In many cases, altered host stromal tissues themselves are critical for many of steps in cancer progression. Stromal endothelial cells and fibroblasts produce many tumor growth factors, which act in paracrine loops. In addition, components of the host tissue matrix and plasma proteins also help promote or inhibit tumor growth. These topics have been extensively reviewed.

A large number of targeted therapies for cancer are also in various stages of clinical development. Due to the likely minimal toxicity and only modest single agent activity of these agents, determining the optimal dose and schedule for these agents will depend upon the identification of biomarkers that can demonstrate proof of target inhibition and/or characterize the downstream consequences of this inhibition.

Despite often robust and durable clinical responses, essentially all patients treated with bevacizumab progress, implying primary or acquired resistance, or both. Treatment related changes in VEGF ligands and receptors have been reported in response to anti-VEGF therapy in preclinical models. Treatment related changes have also been noted for many additional angiogenic factors, including PDGF, bFGF, and IGF, all of which have been shown to potentially mediate sensitivity and resistance to anti-VEGF therapy. Despite the known importance of numerous angiogenic factors in both preclinical models and in patients, there have not yet been a broad and systematic evaluation of either baseline or treatment related changes of multiple angiogenic factors in response to bevacizumab. Similar information is also lacking for essentially all targeted therapies.

Biomarkers to better understand the mechanisms of action, primary and acquired resistance, and toxicity of these agents are urgently needed. The topic has been extensively reviewed and is considered a priority by the NCI. The need for such biomarkers is critical given the increasing number of permutations of targeted therapeutics and the need for biomarkers to guide patient and treatment selection both in clinical trials and in general use of anti-cancer therapy. Assay optimization and defining expected values of each marker or panel of markers is critical before use of such assays in large therapeutic clinical trials designed to target specific patient populations. In addition, understanding the biology and regulation of biomarkers related to tumor growth and tumor angiogenesis is also important. Most candidate biomarkers are themselves cellular growth factors, and are involved in not only tumor promotion and growth, but also in normal growth and development and in normal and abnormal tissues responses to injury. The primary purpose of the proposed project is to help refine new biomarkers and new and evolving technologies to assess them.

ELIGIBILITY:
Inclusion Criteria:

LOCAL (Raleigh-Durham, Chapel Hill) candidates only!!!

* Age >18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects may not have major medical or other conditions that might affect the study assays: major surgery or trauma in the past six months, known current pregnancy, diabetes, history of coagulation abnormalities.
* Subjects may not be receiving any investigational agents.
* Subjects may not be taking medications that are likely to significantly affect wound healing or clotting (eg steroids, anti-coagulants, hormonal contraceptives), aspirin > 325mg/d or other NSAID > once per day, birth control pills or other hormonal contraceptives.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients and patients on combination antiretroviral therapy are ineligible because of the potential for alterations in normal wound healing responses. In addition, subjects who currently have a malignancy or have had malignant disease in the past 5 years are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To refine techniques needed to describe the expected values and variability of multiple angiogenic and tumor growth factor levels in blood and urine, using ELISA and other evolving protein and gene expression and cell capture technologies. | 14 days

SECONDARY OUTCOMES:
To describe the expected values and variability of multiple angiogenic and tumor growth factor levels in blood and urine, including VEGF, bFGF, PDGF, PDEGF, TGFβ, TSP1, and MMP2 and MMP9. Other angiogenic and tumor growth factors may also be evaluated. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Herb Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States